CLINICAL TRIAL: NCT00293215
Title: Phase I Biodistribution Study of 111-Indium-CMD-193 in Patients With Advanced Tumours Expressing the Lewis-Y Antigen
Brief Title: Biodistribution Study of CMD-193 in Patients With Advanced Tumours Expressing the Lewis-Y Antigen
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Abnormal distribution and lack of tumor targeting were observed.
Sponsor: Ludwig Institute for Cancer Research (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LUD2004-015
Record Dates: First submitted 2006-02-15; First posted 2006-02-17 (Estimated); Results first posted 2020-08-10 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (1.0 mg/m^2) (Experimental): Subjects received 111-In-CMD-193 on Day 1 of Cycle 1. Subjects received CMD-193 at a dose of 1.0 mg/m^2 on Day 1 of subsequent 21-day cycles.
  Interventions: Drug: 111-Indium-CMD-193; Drug: CMD-193
- Cohort 2 (2.6 mg/m^2) (Experimental): Subjects received 111-In-CMD-193 on Day 1 of Cycle 1. Subjects received CMD-193 at a dose of 2.6 mg/m^2 on Day 1 of subsequent 21-day cycles.
  Interventions: Drug: 111-Indium-CMD-193; Drug: CMD-193

INTERVENTIONS:
Drug: 111-Indium-CMD-193 — 111-In-CMD-193 (3-7 mCi) was administered as an IV infusion over 60 (± 5) minutes.
Drug: CMD-193 — CMD-193 was administered as an IV infusion over 60 (± 5) minutes.

SUMMARY:
This was a Phase 1 dose-escalation study of CMD-193, a humanized monoclonal antibody linked to the toxin calicheamicin, in subjects with advanced tumors expressing the Lewis-Y antigen. The primary study objective was to determine the biodistribution and pharmacokinetics (PK) of 111-In-CMD-193 (i.e., CMD-193 tagged with a small amount of radioactive Indium [111-In]), with secondary objectives of determining changes in tumor metabolism and describing the antitumor responses to CMD-193.

DETAILED DESCRIPTION:
Subjects received a single infusion of 111-In-CMD-193 on Day 1. Collection of blood for PK and whole body gamma camera imaging for assessment of biodistribution and tumor uptake were performed on Days 1, 2, 3 or 4, 5 or 6, and 7 or 8 following the 111-In-CMD-193 infusion. Subjects were evaluated for safety for 3 hours post-infusion on Day 1 of each cycle, with subsequent safety assessments performed on Days 8 and 15. Blood for human anti-human antibody (HAHA) response was collected pre-infusion, prior to each subsequent cycle (every 3 weeks) and at study discontinuation.

CMD-193 was administered on Day 1 of each subsequent 21-day cycle as a 60 (± 5) minute intravenous (IV) infusion at a dose of 1.0 mg/m^2 in Cohort 1 and 2.6 mg/m^2 in Cohort 2. Each subject received up to 6 cycles of CMD-193 (including the initial infusion of 111-In-CMD-193) until disease progression, unacceptable toxicity, or withdrawal of consent. Up to 6 additional cycles of CMD-193 were permitted if approved by the Sponsor in subjects who tolerated CMD-193 treatment and had evidence of response. Pretreatment medications (e.g., paracetamol, promethazine hydrochloride) were to be administered to reduce the incidence and severity of an anticipated infusion syndrome characterized by fever and chills, and less commonly hypotension.

Restaging by computed tomography (CT) scan was performed at the end of Cycles 2, 4, and 6. Assessment of tumor metabolism was performed by positron emission tomography with 18F-labeled fluorodeoxyglucose (18F-FDG-PET) prior to Cycle 1 and at the time of restaging at the end of Cycles 2 and 4.

ELIGIBILITY:
Inclusion criteria:

1. Signed and dated Institutional Review Board (IRB)-approved informed consent before any protocol-specific screening procedures were performed.
2. Histologically confirmed malignant solid tumor that had progressed following standard therapy, or for which no standard effective treatment was available.
3. Tumor expression of Lewis-Y antigen (≥20% tumor cells positive for Lewis-Y by immunohistochemistry assay).
4. Measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST), including the presence of at least one measurable lesion at least 2 cm in size suitable for 18F-FDG PET imaging.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Life expectancy ≥ 18 weeks.
7. Age ≥18 years.
8. Recovery to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) ≤ Grade 1 toxicity from any significant effects of prior surgery, radiation therapy, and cancer therapy (except alopecia).
9. Renal test: serum creatinine ≤ 1.5 x upper limit of normal (ULN).
10. Hepatic tests: alanine aminotransferase (ALT) levels ≤2.5 x ULN and total bilirubin ≤1.5 x ULN.
11. Pancreatic tests: amylase ≤1.5 x ULN and lipase ≤ 1.5 x ULN.
12. Bone marrow tests: absolute neutrophil count (ANC) of ≥1500 mm^3 (≥1.5 x 10^9/L) and platelet count of ≥ 150,000/mm^3 (≥150 x 10^9/L).
13. For women of childbearing potential, a negative serum pregnancy test result no longer than 48 hours before the first dose of CMD-193. A woman of childbearing potential was one who was biologically capable of becoming pregnant. This included women who were using contraceptives or whose sexual partners were either sterile or using contraceptives.
14. All subjects who were not surgically sterile or postmenopausal must have agreed and committed to the use of a reliable method of birth control for the duration of the study and for 28 days after the last dose of CMD-193.
15. Willingness of female subjects to refrain from breastfeeding infants during the study or within 28 days after the last dose of CMD-193.

Exclusion Criteria

1. Chemotherapy, radiation therapy, other cancer therapy, or investigational agents within 21 days of the first dose of CMD-193 (42 days if the previous chemotherapy included nitrosoureas or mitomycin C).
2. Symptomatic or clinically active central nervous system (CNS) metastases. Subjects who had prior treatment with radiotherapy or surgical resection for CNS metastases were permitted if CNS metastases had remained stable and not required any treatment for at least 3 months prior to the first dose of CMD-193.
3. Significant prior allergic reaction to recombinant human or murine proteins.
4. History of cirrhosis, current or chronic hepatitis B or C infections, or other significant active liver disease.
5. Unstable or serious concurrent medical conditions. Examples included, but were not limited to, bleeding gastric ulcers, gastrointestinal bleeding, hepatitis, significant disorders of the immune system (eg, systemic lupus erythematosus), pancreatitis, congestive heart failure, serious active infections (e.g. requiring antibiotics or antiviral agents), unstable angina, recent myocardial infarction (within 6 months of screening), ongoing maintenance therapy for life-threatening ventricular arrhythmia, or uncontrolled major seizure disorder.
6. Other malignancy within 3 years prior to entry into the study, except for treated non-melanoma skin cancer and cervical carcinoma in situ.
7. Any other condition that, in the Investigator's judgment, would have substantially increased the risk associated with the subject's participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2006-02 (Actual); Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: A/Prof. Andrew M Scott, MBBS MD DDU, Principal Investigator — Ludwig Institute for Cancer Research
Locations (2):
- Australia (2):
  - Cancer Care Services, Dept. of Medical Oncology, Royal Brisbane and Women's Hospital, Herston, Queensland
  - Ludwig Institute Tumor Targeting Program, Austin Health, Heidelberg (Melbourne), Victoria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Therasse P, Arbuck SG, Eisenhauer EA, Wanders J, Kaplan RS, Rubinstein L, Verweij J, Van Glabbeke M, van Oosterom AT, Christian MC, Gwyther SG. New guidelines to evaluate the response to treatment in solid tumors. European Organization for Research and Treatment of Cancer, National Cancer Institute of the United States, National Cancer Institute of Canada. J Natl Cancer Inst. 2000 Feb 2;92(3):205-16. doi: 10.1093/jnci/92.3.205. PMID 10655437
- [Background] Young H, Baum R, Cremerius U, Herholz K, Hoekstra O, Lammertsma AA, Pruim J, Price P. Measurement of clinical and subclinical tumour response using [18F]-fluorodeoxyglucose and positron emission tomography: review and 1999 EORTC recommendations. European Organization for Research and Treatment of Cancer (EORTC) PET Study Group. Eur J Cancer. 1999 Dec;35(13):1773-82. doi: 10.1016/s0959-8049(99)00229-4. PMID 10673991
- [Result] Herbertson RA, Tebbutt NC, Lee FT, MacFarlane DJ, Chappell B, Micallef N, Lee ST, Saunder T, Hopkins W, Smyth FE, Wyld DK, Bellen J, Sonnichsen DS, Brechbiel MW, Murone C, Scott AM. Phase I biodistribution and pharmacokinetic study of Lewis Y-targeting immunoconjugate CMD-193 in patients with advanced epithelial cancers. Clin Cancer Res. 2009 Nov 1;15(21):6709-15. doi: 10.1158/1078-0432.CCR-09-0536. Epub 2009 Oct 13. PMID 19825951

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 (1.0 mg/m^2): Subjects received Indium-111 labelled-CMD-193 (111-In-CMD-193) (3-7 mCi) intravenously (IV) on Day 1 of Cycle 1. Subjects received CMD-193 at a dose of 1.0 mg/m^2 IV on Day 1 of subsequent 21-day cycles.
- Cohort 2 (2.6 mg/m^2): Subjects received 111-In-CMD-193 (3-7 mCi) IV on Day 1 of Cycle 1. Subjects received CMD-193 at a dose of 2.6 mg/m^2 IV on Day 1 of subsequent 21-day cycles.
Period: Overall Study
Arm/Group | Cohort 1 (1.0 mg/m^2) | Cohort 2 (2.6 mg/m^2)
Started | 6 | 3
Completed (Completed the study as planned, i.e., received all 6 cycles of CMD-193) | 1 | 0
Not Completed | 5 | 3
Not completed — Progressive disease | 3 | 1
Not completed — Adverse Event | 2 | 2

BASELINE CHARACTERISTICS:
Population: All enrolled subjects.
Groups:
- Cohort 1 (1.0 mg/m^2): Subjects received 111-In-CMD-193 (3-7 mCi) IV on Day 1 of Cycle 1. Subjects received CMD-193 at a dose of 1.0 mg/m^2 IV on Day 1 of subsequent 21-day cycles.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (1.0 mg/m^2) | Cohort 2 (2.6 mg/m^2) | Total
Number analyzed (Participants) | 6 | 3 | 9
Age, Continuous [Median (Full Range); unit: years] | 53 [46 to 71] | 69 [46 to 77] | 53 [46 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 4 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 1 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 6 | 3 | 9
Primary tumor [Count of Participants; unit: Participants]
  Colon carcinoma | 3 | 0 | 3
  Cholangiocarcinoma | 1 | 0 | 1
  Gastric carcinoma | 1 | 1 | 2
  Gastro-esophageal junction carcinoma | 1 | 0 | 1
  Bronchoalveolar carcinoma | 0 | 1 | 1
  Pulmonary adenocarcinoma | 0 | 1 | 1
Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) [Count of Participants; unit: Participants] — PS 0 = Fully active, able to carry on all pre-disease performance without restriction; PS 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; PS 2 = Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours; PS 3 = Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours; PS 4 = Completely disabled; cannot carry on any selfcare; totally confined to bed or chair; PS 5 = Dead
  Participants
    0 | 5 | 1 | 6
    1 | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Summary of 111-In-CMD-193 Biodistribution Based on Gamma Camera Images
Description: Biodistribution data were collected after subjects received a single infusion of 111-In-CMD-193 over 1 hour on Day 1 of Cycle 1. Gamma camera imaging with anterior and posterior whole body scans using conjugate view methodology were performed on Days 1, 2, 3 or 4, 5 or 6, and 7 or 8 following the 111-In-CMD-193 infusion. A standard was included in the field of view at each imaging time point. Single-photon emission computerized tomography (SPECT) imaging of relevant areas of disease were performed on at least one occasion following the 111-In-CMD-193 infusion. Biodistribution analysis was performed by examination of whole body and SPECT images by experienced nuclear medicine physicians.
Time Frame: Up to 8 days
Population: All subjects who received a single infusion of 111-In-CMD-193 on Day 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (1.0 mg/m^2) | Cohort 2 (2.6 mg/m^2)
Number analyzed (Participants) | 6 | 3
Participants
  Initial blood pooling | 6 | 3
  Hepatic uptake by Day 2 persisting to Day 8 | 6 | 3
  Fast blood clearance | 6 | 3
  Tumor uptake | 0 | 0

2. Primary Outcome: Mean Effective Half-life of 111-In-CMD-193 Based on Gamma Camera Images
Description: Gamma camera imaging with anterior and posterior whole body scans using conjugate view methodology were performed on Days 1, 2, 3 or 4, 5 or 6, and 7 or 8 following the 111-In-CMD-193 infusion. Whole body clearance, or biological half-time, was calculated from the whole body anterior and posterior planar images. A region of interest (ROI) was calculated to encompass the whole body, and for each ROI at each time point, the mean counts per pixel per minute was normalized to imaging time point Day 1. From this time-activity curve, an exponential clearance expression was fitted to obtain effective half-time. This was then corrected for the physical half-life of 111-In (67.45 hours) to account for physical decay to obtain the biological half-time.
Time Frame: Up to 8 days
Population: All subjects who received a single infusion of 111-In-CMD-193 on Day 1.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cohort 1 (1.0 mg/m^2) | Cohort 2 (2.6 mg/m^2)
Number analyzed (Participants) | 6 | 3
hours | 47.54 (3.16) | 48.37 (4.03)

3. Primary Outcome: Mean Serum Half-lives of 111-In-CMD-193
Description: During Cycle 1 (111-In-CMD-193 infusion) serum samples for pharmacokinetics were collected on Days 1 (pre-infusion and 1 and 4 hours after the start of the infusion), 3, 8 and 15. Serum obtained from subjects following infusion of 111-In-CMD-193 was aliquoted and counted in a gamma scintillation counter. Duplicate standards prepared from the injected material were counted at each time point with serum samples to enable calculations to be corrected for the isotope physical decay. A 2-compartment IV bolus model with macro-parameters, no lag time and first order elimination (WNL Model 8) was fitted to individual labelled infusions for each subject using un-weighted nonlinear, least squares with WinNonLin version 5.2. T½α and T½β represent half lives of the initial and terminal phases of disposition.
Time Frame: Approximately 15 days (i.e., Days 1, 3, 8, and 15)
Population: All subjects who received a single infusion of 111-In-CMD-193 on Day 1.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cohort 1 (1.0 mg/m^2) | Cohort 2 (2.6 mg/m^2)
Number analyzed (Participants) | 6 | 3
hours
  T½α | 5.47 (1.99) | 3.32 (2.00)
  T½β | 104.42 (37.94) | 99.79 (38.32)

4. Primary Outcome: Mean Volume of Central Compartment of 111-In-CMD-193
Description: During Cycle 1 (111-In-CMD-193 infusion) serum samples for pharmacokinetics were collected on Days 1 (pre-infusion and 1 and 4 hours after the start of the infusion), 3, 8 and 15. Serum obtained from subjects following infusion of 111-In-CMD-193 was aliquoted and counted in a gamma scintillation counter. Duplicate standards prepared from the injected material were counted at each time point with serum samples to enable calculations to be corrected for the isotope physical decay. A 2-compartment IV bolus model with macro-parameters, no lag time and first order elimination (WNL Model 8) was fitted to individual labelled infusions for each subject using un-weighted nonlinear, least squares with WinNonLin version 5.2.
Time Frame: Approximately 15 days (i.e., Days 1, 3, 8, and 15)
Population: All subjects who received a single infusion of 111-In-CMD-193 on Day 1.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Cohort 1 (1.0 mg/m^2) | Cohort 2 (2.6 mg/m^2)
Number analyzed (Participants) | 6 | 3
mL | 4366.18 (586.87) | 3481.31 (704.13)

5. Primary Outcome: Mean Total Serum Clearance of 111-In-CMD-193
Description: as for outcome 4
Time Frame: Approximately 15 days (i.e., Days 1, 3, 8, and 15)
Population: All subjects who received a single infusion of 111-In-CMD-193 on Day 1.
Measure: Mean (Standard Deviation); unit: mL/hr
Arm/Group | Cohort 1 (1.0 mg/m^2) | Cohort 2 (2.6 mg/m^2)
Number analyzed (Participants) | 6 | 3
mL/hr | 130.04 (61.25) | 79.56 (29.67)

6. Primary Outcome: Mean Area Under the Serum Concentration Curve Extrapolated to Infinite Time for 111-In-CMD-193
Description: as for outcome 4
Time Frame: Approximately 15 days (i.e., Days 1, 3, 8, and 15)
Population: All subjects who received a single infusion of 111-In-CMD-193 on Day 1.
Measure: Mean (Standard Deviation); unit: μg*hr/mL
Arm/Group | Cohort 1 (1.0 mg/m^2) | Cohort 2 (2.6 mg/m^2)
Number analyzed (Participants) | 6 | 3
μg*hr/mL | 16.37 (6.13) | 56.45 (17.05)

7. Secondary Outcome: Number of Subjects With Best Tumor Response as Measured by the Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Computed tomography (CT) scans were performed at screening, between Days 15 and 21 of Cycles 2 and 4, and at study completion. Response was assessed using RECIST version 1.0 (Therasse et al, J Natl Cancer Inst 2000; 92:205-16), and all response assessment was performed by a single experienced radiologist. Per RECIST, target lesions are categorized as follows: complete response (CR): disappearance of all target lesions (no evaluable disease); partial response (PR): ≥ 30% decrease in the sum of the longest diameter of target lesions; progressive disease (PD): ≥ 20% increase in the sum of the longest diameter of target lesions; stable disease (SD): small changes that do not meet above criteria.
Time Frame: Up to 4 months
Population: All subjects who received at least 1 dose of study treatment and completed protocol procedures through at least 21 days following their first cycle.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (1.0 mg/m^2) | Cohort 2 (2.6 mg/m^2)
Number analyzed (Participants) | 6 | 2
Participants
  Stable disease | 3 | 2
  Progressive disease | 3 | 0

8. Secondary Outcome: Number of Subjects With Best Metabolic Tumor Response by European Organisation for Research and Treatment of Cancer (EORTC) Guidelines at End of Study
Description: Positron emission tomography with 18F-labeled fluorodeoxyglucose (18F-FDG-PET) was done at screening and between Days 15-21 of Cycles 2 and 4 or at study completion. Metabolic response was calculated using the target lesion with the greatest baseline standardized uptake value (SUV) and categorized per EORTC guidelines (Young et al. Eur J Cancer 1999;35:1773-82): progressive metabolic disease was an increase in 18F-FDG tumor maximum SUV (SUVmax) of > 25% within the tumor ROI determined on baseline scans, visible increase in 18F-FDG tumor uptake (>20% in the longest dimension) or new 18F-FDG uptake in metastatic lesions. Stable metabolic disease was an increase in tumor 18F-FDG SUVmax of < 25% or decrease of < 15% and no visible increase in 18F-FDG tumor uptake (>20% in the longest dimension). Partial metabolic response was a reduction of 15-25% in tumor 18F-FDG SUVmax after 1 cycle and > 25% after > 1 cycle (reduced tumor 18F-FDG uptake was not required).
Time Frame: Up to 4 months
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (1.0 mg/m^2) | Cohort 2 (2.6 mg/m^2)
Number analyzed (Participants) | 6 | 2
Participants
  Partial metabolic response | 1 | 0
  Stable metabolic disease | 2 | 1
  Progressive metabolic disease | 3 | 1

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) occurring between the first dose of study treatment and the off-study date (i.e., up to 4 months) were documented, regardless of the causal relationship to study drug.
Description: AE documentation included onset/resolution dates, severity using the NCI CTCAE (version 3.0), seriousness, relationship to study drug, study drug action taken, treatment, and outcome.
Arm/Group | Cohort 1 (1.0 mg/m^2) | Cohort 2 (2.6 mg/m^2)
All-Cause Mortality (participants affected / at risk) | 0/6 | 1/3
Serious Adverse Events (participants affected / at risk) | 1/6 | 1/3
Other Adverse Events (participants affected / at risk) | 6/6 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (1.0 mg/m^2) (N=6) | Cohort 2 (2.6 mg/m^2) (N=3)
Biliary sepsis (Infections and infestations) | 1 | 0
Malignant pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (1.0 mg/m^2) (N=6) | Cohort 2 (2.6 mg/m^2) (N=3)
Anaemia (Blood and lymphatic system disorders) | 5 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 2
Neutropenia (Blood and lymphatic system disorders) | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 2
Gastroesophageal reflux (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 5 | 2
Vomiting (Gastrointestinal disorders) | 2 | 2
Ankle oedema (General disorders) | 3 | 0
Flushing (General disorders) | 1 | 0
Lethargy (General disorders) | 6 | 0
Alkaline phosphatase increased (Investigations) | 4 | 1
Anorexia (Metabolism and nutrition disorders) | 5 | 3
Dizziness (Nervous system disorders) | 1 | 1
Vasovagal symptoms (Nervous system disorders) | 1 | 0
Bruising (Skin and subcutaneous tissue disorders) | 1 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Epigastric pain (Gastrointestinal disorders) | 1 | 0
Right upper quadrant pain (Gastrointestinal disorders) | 1 | 1
Cold symptoms (Infections and infestations) | 1 | 0
Weight loss (Investigations) | 1 | 1
Headache (Nervous system disorders) | 1 | 1
Sebaceous cyst (Skin and subcutaneous tissue disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 0
Flu-like symptoms (General disorders) | 2 | 0
Oedematous feet (General disorders) | 1 | 0
Pitting oedema (General disorders) | 2 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 3
Alanine aminotransferase increased (Investigations) | 3 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 2
Gamma-glutamyltransferase increased (Investigations) | 2 | 1
Lactate dehydrogenase increased (Investigations) | 1 | 0
Lipase increased (Investigations) | 3 | 0
Proteins serum plasma low (Investigations) | 1 | 1
Discolouration skin (Skin and subcutaneous tissue disorders) | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 3 | 1
Epigastric discomfort (Gastrointestinal disorders) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Abdominal crampy pains (Gastrointestinal disorders) | 1 | 0
Tenderness epigastric (Gastrointestinal disorders) | 1 | 0
Head cold (Infections and infestations) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in hip (Musculoskeletal and connective tissue disorders) | 1 | 0
Weakness in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Paresthesia of fingers (Nervous system disorders) | 1 | 0
Confusion (Psychiatric disorders) | 1 | 0
Hallucinations (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 0
Abdominal bloating (Gastrointestinal disorders) | 1 | 0
Abdominal noises (Gastrointestinal disorders) | 1 | 0
Amylase increased (Investigations) | 0 | 1
Chloride low (Investigations) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Crackles lung (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Runny nose (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Neutrophilia (Blood and lymphatic system disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Following an interim review of primary endpoint data, the study was terminated early on the basis of abnormal distribution and lack of tumor targeting in both dose cohorts.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less